CLINICAL TRIAL: NCT03302559
Title: Assessing the Cosmetic Changes in the Facial Skin Utilizing Non-Invasive In Vivo Skin Imaging Instrumentation After Use of a Topical Retinoid Product In Subjects With Moderate to Severe Photodamage
Brief Title: Study to Assess the Cosmetic Changes in the Facial Skin After Use of a Topical Retinoid Product in Participants With Moderate to Severe Photodamage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRIC17-RET05
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Skin Care
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Retinol Complex 0.5 (Experimental): During a 2-week washout period the participant used a basic skin care regimen (SkinMedica facial cleanser in the morning and in the evening, Cetaphil Fragrance Free Moisturizing Lotion in the morning and in the evening and SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen in the morning and as needed), followed by the same basic skin care regimen plus SkinMedica Retinol Complex 0.5 applied topically to the face in the evening for 12 Weeks. Assessments of the participant's facial skin were made utilizing investigator clinical grading, digital photography, a spectrophotometer and in vivo skin imaging.
  Interventions: Other: Retinol Complex 0.5; Other: Facial cleanser; Other: Moisturizing lotion; Other: Sunscreen; Device: Skin Imaging

INTERVENTIONS:
Other: Retinol Complex 0.5 — Retinol Complex 0.5 topically in the evening.
  Other Names: SkinMedica Retinol Complex 0.5
Other: Facial cleanser — Facial cleanser in the morning and in the evening.
  Other Names: SkinMedica Facial Cleanser
Other: Moisturizing lotion — Fragrance free moisturizing lotion in the morning and in the evening.
  Other Names: Cetaphil Fragrance Free Moisturizing Lotion
Other: Sunscreen — Sunscreen broad spectrum sun protection factor (SPF) 35 topically in the morning and as needed.
  Other Names: SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35
Device: Skin Imaging — Non-invasive in vivo skin imaging will be taken with the VivoSight Dx Optical Coherence Tomography (OCT) and VivaScope 1500

SUMMARY:
This study will assess the cosmetic changes of a cosmetic topical retinoid product in participants with moderate to severe photodamage utilizing non-invasive in vivo skin imaging instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Fitzpatrick skin type I-IV
* Presence of moderate to severe facial photodamage
* Participants taking hormone replacement or hormones for birth control, willing to stop or change this medication for the duration of the study
* Willingness to cleanse the face and remove all makeup at least 15 minutes prior to each scheduled clinic visit
* Willingness to not use any other products, including self-tanners on their facial skin during the study
* Willingness to avoid as much as possible, direct and prolonged sun exposure for the duration of the study (including tanning beds), especially from 10 AM to 2 PM. Participants are asked to wear protective clothing prior to and during exposure.

Exclusion Criteria:

* Individuals with active symptoms of allergy, cold sore or warts, active psoriasis or eczema, rosacea, sunburn, open wounds, neurotic excoriations, excessive scarring, tattoos, or other skin conditions in the test areas that would interfere with the assessments of this study
* Individuals who are nursing, pregnant, or planning to become pregnant during the study
* Individuals with uncontrolled disease such as diabetes, hypertension, hyper or hypothyroidism, active hepatitis, immune deficiency, or autoimmune
* Individuals who have a pre-existing or dormant dermatologic condition (e.g., psoriasis, atopic dermatitis, rosacea, skin cancer, etc.)
* Individuals who require electrolysis, waxing, or use depilatories on the face during the study
* Chemical peel or microdermabrasion within 4 weeks of study start
* Retin-A®, Retin-A Micro®, Renova®, Avita®,Tazorac®, Avage® or Differin® or other similar prescription drugs within 3 months of study start
* Cosmetic injections (filler and/or toxins, i.e. Juvederm, Radiesse, Botox, etc.), non-ablative laser or fractional laser resurfacing
* Accutane® or other oral retinoid, Ablative procedures (i.e. laser, chemical, cosmetic surgeries) within 12 months of study start
* Participants who have planned surgeries or procedures.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Goberdhan, B.A., Principal Investigator — Allergan
Locations (1):
- SkinMedica Clinical Research and Innovation Center, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retinol Complex 0.5
Started | 29
Completed | 23
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrew Consent | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all enrolled participants who applied the test product and completed one follow-up visit after test product was initiated.
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11
  Hispanic | 3
  Asian | 8
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Photodamage Score
Description: The investigator assessed the participant's overall photodamage using a 10-point scale where None (0)= Facial skin is smooth to the touch, without significant fine/coarse line or skin tone unevenness in any areas (periocular, cheeks, forehead and perioral areas) to Severe (7 to 9)= Facial skin shows 3 or more areas (periocular, cheeks, forehead and perioral areas) of significant roughness, skin tone unevenness (red/brown), or fine/coarse lines at Baseline and Week 12. A decrease in score indicates improvement. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT Population included all enrolled participants who applied the test product and completed one follow-up visit after test product was initiated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Baseline (BL) | 5.6 (0.9)
  Change from BL at Week 12 | -0.8 (0.5)
Statistical Analysis 1: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12; Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p < 0.001, Paired t-test — Statistical significance is defined as a p-value ≤0.05

2. Primary Outcome: Change From Baseline in Appearance of Fine Lines/Wrinkles Score (Forehead, Periocular, Cheeks and Perioral Areas Individually Assessed)
Description: The investigator assessed the participant's appearance of fine lines/wrinkles using a 10-point scale where None (0)= No fine lines/wrinkles present; skin looks completely smooth and wrinkle-free to Severe (7 to 9)= Many coarse lines/wrinkles densely packed together in the treatment area (forehead, periocular, cheeks and perioral areas) at Baseline and Week 12. A decrease in score indicates improvement. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Baseline (Forehead) | 3.4 (1.5)
  Change from BL at Week 12 (Forehead) | -0.8 (1.2)
  Baseline (Periocular) | 4.7 (1.5)
  Change from BL at Week 12 (Periocular) | -1.0 (1.8)
  Baseline (Cheeks) | 3.6 (1.5)
  Change from BL at Week 12 (Cheeks) | -1.1 (1.3)
  Baseline (Perioral) | 4.0 (1.6)
  Change from BL at Week 12 (Perioral) | -0.9 (1.2)
Statistical Analysis 1: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Forehead); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.005, Paired t-test — Statistical significance is defined as a p-value ≤0.05
Statistical Analysis 2: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Periocular); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.02, Paired t-test — Statistical significance is defined as a p-value ≤0.05
Statistical Analysis 3: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Cheeks); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.0006, Paired t-test — Statistical significance is defined as a p-value ≤0.05
Statistical Analysis 4: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Perioral); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.001, Paired t-test — Statistical significance is defined as a p-value ≤0.05

3. Primary Outcome: Change From Baseline in Appearance of Coarse Lines/Wrinkles Score (Forehead, Periocular, Cheeks and Perioral Areas Individually Assessed)
Description: The investigator assessed the participant's appearance of coarse lines/wrinkles using a 10-point scale where None (0)= No coarse lines/wrinkles present; skin looks completely smooth and wrinkle-free to Severe (7 to 9)= Many coarse lines/wrinkles densely packed together in the treatment area (forehead, periocular, cheeks and perioral areas) at Baseline and Week 12. A decrease in score indicates improvement. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT Population included all enrolled participants who applied study treatment and completed one follow-up visit after test product was initiated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Baseline (Forehead) | 4.9 (1.4)
  Change from BL at Week 12 (Forehead) | -0.6 (1.1)
  Baseline (Periocular) | 6.0 (1.2)
  Change from Baseline at Week 12 (Periocular) | -0.7 (1.0)
  Baseline (Cheeks) | 3.5 (2.4)
  Change from Baseline at Week 12 (Cheeks) | -1.1 (1.1)
  Baseline (Perioral) | 4.4 (1.9)
  Change from BL at Week 12 (Perioral) | -0.2 (1.2)
Statistical Analysis 1: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Forehead); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.02, Paired t-test — Statistical significance is defined as a p-value ≤0.05
Statistical Analysis 2: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Periocular); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.006, Paired t-test — Statistical significance is defined as a p-value ≤0.05
Statistical Analysis 3: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Cheeks); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p < 0.001, Paired t-test — Statistical significance is defined as a p-value ≤0.05
Statistical Analysis 4: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Perioral); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.5, Paired t-test — Statistical significance is defined as a p-value ≤0.05

4. Primary Outcome: Change From Baseline in Tactile Roughness Score
Description: The investigator assessed the participant's tactile roughness in the entire face using a 10-point scale where None (0)= No roughness of the treatment area; skin is completely smooth and pliable to Severe (7 to 9)= Marked roughness of the treatment area associated with stiff feeling at Baseline and Week 12. A decrease in score indicates improvement. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Baseline | 4.0 (1.7)
  Change from BL at Week 12 | -1.1 (1.6)
Statistical Analysis 1: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12; Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.002, Paired t-test — Statistical significance is defined as a p-value ≤0.05

5. Secondary Outcome: Change From Baseline in Skin Roughness Score Using the Allergan Skin Roughness Visual Scale
Description: The investigator assessed the participant's skin roughness using the Allergan Skin Roughness Visual 5-Point Scale where None (0)= Smooth visual skin texture to Extreme (4)= Extremely coarse visual skin texture, crosshatched deep creases; extreme elastosis at Baseline and Week 12. A decrease in score indicates improvement. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT Population included all enrolled participant who applied study treatment and completed one follow-up visit after test product was initiated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Baseline | 1.8 (1.1)
  Change from BL at Week 12 | -0.5 (0.6)
Statistical Analysis 1: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12; Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.0008, Paired t-test — Statistical significance is defined as a p-value ≤0.05

6. Secondary Outcome: Change From Baseline in Appearance of Fine Lines Score Using the Allergan Fine Lines Visual Scale
Description: The investigator assessed the participant's fine lines using the Allergan Fine Lines Visual 5-Point Scale where None (0)= No fine lines to Diffuse (4)= Diffuse superficial lines; crosshatching at Baseline and Week 12. A decrease in score indicates improvement. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Baseline | 4.0 (1.7)
  Change from BL at Week 12 | -0.3 (0.6)
Statistical Analysis 1: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12; Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.02, Paired t-test — Statistical significance is defined as a p-value ≤0.05

7. Secondary Outcome: Investigator's Global Improvement Assessment for Overall Photodamage
Description: The investigator assessed the global improvement in the participant's overall photodamage compared to Baseline using a 5-point scale where None (0)= No change or worsening to Complete (4)= Almost complete improvement of the condition with a trace of signs/symptoms remaining (approximately 95% or better overall improvement).
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale | 1.5 (0.7)

8. Secondary Outcome: Investigator's Global Improvement Assessment for the Appearance of Fine Lines/Wrinkles (Forehead, Periocular, Cheeks, Perioral Areas Individually Assessed)
Description: The investigator assessed the global improvement in the participant's overall appearance of fine lines/wrinkles compared to Baseline using a 5-point scale where None (0)= No change or worsening to Complete (4)= Complete clearing in the appearance of fine lines/wrinkles (approximately 95% or better overall improvement).
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Week 12 (Forehead) | 1.1 (0.6)
  Week 12 (Periocular) | 1.6 (0.9)
  Week 12 (Cheeks) | 1.3 (0.6)
  Week 12 (Perioral) | 1.2 (0.7)

9. Secondary Outcome: Investigator's Global Improvement Assessment for the Appearance of Coarse Lines/Wrinkles (Forehead, Periocular, Cheeks, Perioral Areas Individually Assessed)
Description: The investigator assessed the global improvement in the participant's overall appearance of coarse lines/wrinkles compared to Baseline using a 5-point scale where None (0)= No change or worsening to Complete (4)= Complete clearing in the appearance of coarse lines/wrinkles (approximately 95% or better overall improvement).
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Week 12 (Forehead) | 0.8 (0.8)
  Week 12 (Periocular) | 1.6 (0.8)
  Week 12 (Cheeks) | 0.9 (0.8)
  Week 12 (Perioral) | 0.8 (0.8)

10. Secondary Outcome: Investigator's Global Improvement Assessment for Tactile Roughness
Description: The investigator assessed the global improvement in the participant's overall tactile roughness compared to Baseline using a 5-point scale where None (0)= No change or worsening to Complete (4)= Complete clearing in the appearance of tactile roughness (approximately 95% or better overall improvement).
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale | 1.3 (1.1)

11. Secondary Outcome: Change From Baseline in Spectrophotometer L* Value (a Measurement of Skin Brightness)
Description: Triplicate spectrophotometer readings were taken of the participant's face (Normal Skin and Target Lesions) at Baseline and Week 12. L* value scores range from 0=black to 100=white. An increase in the spectrophotometer L* values indicates improvement. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT Population included all enrolled participants who applied study treatment and completed one follow-up visit after test product was initiated. Number analyzed is the number of participants with data available at the given time-point for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Retinol Complex 0.5
Number analyzed (Participants) | 23
score on a scale
  Baseline (Normal Skin) | 62.0 (3.7)
  Change from BL at Week 12 (Normal Skin) | 0.3 (1.8)
  Baseline (Target Lesion) | 57.8 (5.7)
  Change from BL at Week 12 (Target Lesion): number analyzed (Participants) | 16
  Change from BL at Week 12 (Target Lesion) | 0.3 (1.7)
Statistical Analysis 1: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Normal Skin); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.3, Paired t-test — Statistical significance is defined as a p-value ≤0.05
Statistical Analysis 2: Comparison: Retinol Complex 0.5; Change from Baseline at Week 12 (Target Lesion); Test type: Other — Testing hypothesis is that the mean change from baseline is zero; p = 0.4, Paired t-test — Statistical significance is defined as a p-value ≤0.05

ADVERSE EVENTS:
Time Frame: First study treatment application up to 12 weeks
Description: Enrolled Population was used to determine the number of participants at risk for All-Cause Mortality. Safety Population, all enrolled participants who applied the test product, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Retinol Complex 0.5
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 12/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Retinol Complex 0.5 (N=23)
Burning sensation (Skin and subcutaneous tissue disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT03302559/Prot_SAP_000.pdf